CLINICAL TRIAL: NCT05582967
Title: An Observational Cohort Study of People Attending the ED With Symptoms of Acute Aortic Syndrome (AAS)
Brief Title: The DAShED (Diagnosis of Aortic Syndrome in the ED) Study
Acronym: DAShED
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Collaborators: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC22083; 22/PR/0807 (Other: Research Ethics Committee); 315948 (Other: IRAS)
Record Dates: First submitted 2022-10-10; First posted 2022-10-17 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2022-10

CONDITIONS: Aortic Dissection
Keywords: Aortic Dissection; Diagnostic accuracy; Aorta; Emergency; Diagnosis
MeSH Terms: conditions — Aortic Dissection; Emergencies; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Completion of focused Electronic Case Report Form — All patients will have a focussed Electronic Case Report Form completed collecting information around Presenting complaint, Past Medical History, Family History, Physical Examination findings, and Investigations.

SUMMARY:
Acute aortic syndrome (AAS) is a life-threatening emergency condition affecting the upper aorta affecting ~4000 people in the (United Kingdom; UK) a year with an ED misdiagnosis rate as high as 38%. Previous research has identified several strategies combining clinical probability scoring with blood tests (D-Dimer) to rule out the condition but when applied to a large population (ED) with relatively low numbers of actual cases, these result in a high rate of computed tomographic angiography (CTA) scanning. Current guidelines reflect the uncertainty of existing evidence.

This study, the first phase of three, aims to describe the characteristics of ED attendances with possible AAS, to determine the service implications of using different diagnostic strategies and inform future research. The investigators plan to recruit all ED attendances with possible AAS over a 1-4 week period. The investigators plan a prospective and retrospective approach to data collection adopting a waived-consent strategy with endpoint measures describing the characteristics of patients presenting with possible AAS.

DETAILED DESCRIPTION:
AAS is a life-threatening emergency condition which presents to the ED. Around 4,000 people suffer per year in the UK [1], many not receiving timely diagnosis and treatment. 25% of patients are not diagnosed until 24 hours after arriving in the ED due to the varied nature of presentation [2]. Chest pain is the most common presenting symptom of AAS (80%) although back pain (40%) and abdominal pain are not uncommon [1]. These symptoms account for over 2 million ED attendances per year in England [National Health Service; NHS Digital A&E 2021] and are overwhelmingly due to causes other than AAS. The estimated incidence of AAS is 1 in every 980 ED attendances with atraumatic chest pain [3], thus creating a substantial diagnostic challenge.

Prognosis is best when patients are treated early, and mortality increases 2% per hour of delay. [4] The misdiagnosis rate during the initial ED visit for AAS is estimated to be between 1 in 3 to 1 in 7 AASs [5], leading to worse outcomes [6,7] whilst CTA over testing leads to diagnostic yields as low as 2-3%. [2,8]. CTA scanning of the aorta has high sensitivity and specificity for diagnosing AAS, but an unrestricted CT strategy will incur significant costs, has ionising radiation risks, resource implications, CT delays for non-AAS patients and the burden of 'incidentalomas'.

Clinicians therefore need to use CTA selectively but there is no validated scoring system to help this decision. Several have been proposed [1, 9-14] including the ADD-RS score, the Canadian clinical practice guideline Clinical Decision Aid [13], the AORTAs score [14] and the Sheffield score [unpublished]. D-Dimer has been suggested as a rule-out biomarker in low pre-test probability patients (95-98% sensitivity) [15,16] and has been incorporated into the Aortic Dissection Detection-Risk Stratification (ADD-RS) score to reduce CTA rate in low pre-test probability patients. None have been studied in truly undifferentiated ED populations, or in the UK where CTA threshold is different compared to North America. It is currently unclear whether any have sufficient sensitivity to be acceptable to clinicians, which is the most accurate, and whether they are likely to lead to CTA and D-Dimer over testing. Assessment of CTA rate and CT positivity has also not previously been studied. The Royal College of Emergency Medicine has recently released a national guideline advocating any patient with an ADD-RS score of >=1 (no D-dimer incorporated) should have a CT aorta performed (unless other cause for symptoms identified and evidenced). The recommendation is not based on UK-validated clinical evidence, however, and clinical impacts of the recommendation are yet to be seen.

In view of these diagnostic challenges, the investigators aim in our programme of work to ultimately to assess which of the four aforementioned clinical decision tools is most effective, assess external validity, and assess clinical impact. This study (Phase 1; DAShED) will involve prospective data collection on all characteristics of four different risk scores, in addition to evaluation of patient characteristics, potential CT aorta rates with different strategies, and enrolment rates at participating sites. This will inform Phase 2, which will involve full interventional external validation study of the decision aid(s) selected in Phase 1 (including biomarker collection); the main objective being to select the score to subject to assessment of clinical impact (intervention step-wedge trial) in Phase 3.

This is an observational cohort study of all people attending the ED with symptoms of possible AAS, including new-onset chest, back or abdominal pain, syncope or symptoms related to malperfusion.

ELIGIBILITY:
Inclusion Criteria:

* People attending the ED with symptoms of AAS, including those with new-onset chest, back or abdominal pain, syncope or symptoms related to malperfusion.
* ≥16 years old

Exclusion Criteria:

* No symptoms of AAS.
* <16 years old

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All people attending the Emergency Department (ED) with symptoms of possible AAS, including new-onset chest, back or abdominal pain, syncope or symptoms related to malperfusion.
Sampling Method: Non-Probability Sample
Enrollment: 5548 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-01-21 (Actual); Study Completion 2023-01-21 (Actual)

PRIMARY OUTCOMES:
Enrolment rate at each participating site | 30 days
  Number of participants during study period enrolled
Proportion of patients in whom the ED clinician thinks Acute Aortic Syndrome (AAS) is a possible differential who have confirmed AAS | 30 days
  Proportion of patients in whom the ED clinician thinks Acute Aortic Syndrome (AAS) is a possible differential who have confirmed AAS
Proportion of patients in whom ED clinician considers AAS NOT a possible differential who had confirmed AAS | 30 days
  Proportion of patients in whom ED clinician considers AAS NOT a possible differential who had confirmed AAS
Number of AAS patients not enrolled due to lack of clinical/research support | 30 days
  Number of AAS patients not enrolled due to lack of clinical/research support
CT angiogram (CTA) ordering and positivity rate | 30 days
  Number of CT angiograms ordered and the proportion that are positive scans
Test characteristics of clinical acumen | 30 days
  Test characteristics of clinical acumen (i.e. sensitivity, specificity, positive predictive value, negative predictive value)
Test characteristics of ADD-RS (Aortic Dissection Detection-Risk Score) | 30 days
  Test characteristics of Aortic Dissection Detection-Risk Score (i.e. sensitivity, specificity, positive predictive value, negative predictive value)
Test characteristics Aorta score | 30 days
  Test characteristics of Aorta score (i.e. sensitivity, specificity, positive predictive value, negative predictive value)
Test characteristics of Canadian guideline score | 30 days
  Test characteristics of Canadian guideline score (i.e. sensitivity, specificity, positive predictive value, negative predictive value)
Test characteristics of Sheffield AAS decision rule | 30 days
  Test characteristics of Sheffield AAS decision rule (i.e. sensitivity, specificity, positive predictive value, negative predictive value)
Test characteristics of D-dimer | 30 days
  Test characteristics of D-dimer (i.e. sensitivity, specificity, positive predictive value, negative predictive value)
Median time from hospital presentation to imaging diagnosis and median time from symptom onset to hospital presentation (hours) | 30 days
  Median time from hospital presentation to imaging diagnosis and median time from symptom onset to hospital presentation (hours)
30-day mortality in proven AAS | 30 days
  30-day mortality in proven AAS
Proportion of alternative diagnoses found on CTA and final hospital diagnosis | 30 days
  Proportion of alternative diagnoses found on CTA and final hospital diagnosis
Number of patients not able to be enrolled with reason why not enrolled | 30 days
  Number of patients not able to be enrolled with reason why not enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Rachel McLatchie, Principal Investigator — Accord Clinical Research
Locations (25):
- United Kingdom (25):
  - Royal United Hospital, Bath
  - Bristol Royal Infirmary, Bristol
  - North Bristol NHS Trust, Bristol
  - Addenbrookes hospital, Cambridge
  - Royal Infirmary of Edinburgh, Edinburgh
  - St Johns Hospital, Edinburgh
  - Frimley Health, Frimley
  - Queen Elizabeth University Hospital, Glasgow
  - Royal Alexandra Hospital, Glasgow
  - James Paget University Hospital, Great Yarmouth
  - Harrogate, Harrogate
  - Raigmore, Inverness
  - Queen Elizabeth Hospital NHS Foundation Trust, Kings Lynn
  - Victoria Hospital, Kirkcaldy
  - Lewisham and Greenwich NHS Trust, Lewisham
  - Luton & Dunstable University Hospital, Luton
  - Wythenshawe Hospital, Manchester
  - Milton Keynes Universoty Hospital NHS Foundation Trust, Milton Keynes
  - Royal Victoria Infirmary, Newcastle
  - Royal Oldham Hospital, Oldham
  - John Radcliffe Hospital, Oxford
  - Royal Glamorgan Hospital, Pont-y-clun
  - Royal Berkshire NHS Foundation Trust, Reading
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Wexham Park, Slough

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared on request

REFERENCES:
- [Derived] McLatchie R, Reed MJ, Freeman N, Parker RA, Wilson S, Goodacre S, Cowan A, Boyle J, Clarke B, Clarke E; DAShED investigators. Diagnosis of Acute Aortic Syndrome in the Emergency Department (DAShED) study: an observational cohort study of people attending the emergency department with symptoms consistent with acute aortic syndrome. Emerg Med J. 2024 Feb 20;41(3):136-144. doi: 10.1136/emermed-2023-213266. PMID 37945311
- See also: Study website — http://www.emergeresearch.org/trial/dashed/